CLINICAL TRIAL: NCT02292563
Title: Can Experienced Endoscopy Nurse Participation During Screening Colonoscopy Increase Polyp and Adenoma Detection Rate?:A Prospective Randomized Trial
Brief Title: The Impact of Experienced Endoscopy Nurse Participation on Polyp and Adenoma Detection During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Lei Xu, M.D, Ningbo No. 1 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBYY2014001
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2015-10

CONDITIONS: Polyp; Adenoma
Keywords: Nurse; Colonoscopy; Polyp; Adenoma;
MeSH Terms: conditions — Polyps; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- endoscopist only (Experimental): Single inspection by endoscopist during colonoscopy
  Interventions: Procedure: Colonoscopist only; Procedure: Experienced Endoscopy Nurse Participation
- nurse participation (Experimental): Dual inspection by both an endoscopist and an experienced nurse during colonoscopy
  Interventions: Procedure: Colonoscopist only; Procedure: Experienced Endoscopy Nurse Participation

INTERVENTIONS:
Procedure: Colonoscopist only — Only Colonosopist Observe during Colonoscopy (single observer)
Procedure: Experienced Endoscopy Nurse Participation — Experienced Endoscopy Nurse Participation Observation during Colonoscopy (Both endoscopist and endoscopic nurse observe)

SUMMARY:
The purpose of this study is to determine whether experienced endoscopy nurse participation during screening colonoscopy could increase polyp and adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* age 40-70 average risk screening colonoscopy

Exclusion Criteria:

* GI Bleeding ;
* history of colorectal surgery ;
* inflammatory bowel disease ;
* colorectal cancer,or polyposis syndrome

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate | 1.5 year
adenoma detection rate | 1.5 year

SECONDARY OUTCOMES:
Advanced polyp detection rate | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: XIAOYUN DING, M.D, Study Director — Ningbo No. 1 Hospital
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Wang W, Xu L, Bao Z, Sun L, Hu C, Zhou F, Xu L, Shi D. Differences with experienced nurse assistance during colonoscopy in detecting polyp and adenoma: a randomized clinical trial. Int J Colorectal Dis. 2018 May;33(5):561-566. doi: 10.1007/s00384-018-3003-0. Epub 2018 Mar 14. PMID 29541895